CLINICAL TRIAL: NCT05188651
Title: Effect of FFP2 Masks on Peripheral Oxygen Saturation and Pulse Rate During the COVID-19 Pandemic
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Anna Alessandri Bonetti, PhD student, Institute of dental clinic and maxillofacial surgery, Catholic University of the Sacred Heart
Other Study IDs: 4235
Record Dates: First submitted 2022-01-10; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Hypoxia; Hypercapnia; COVID-19 Pandemic
MeSH Terms: conditions — Hypoxia; Hypercapnia; COVID-19 | interventions — Masks

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- dental professionals wearing FFP2/N95 masks
  Interventions: Behavioral: face masks
- dental professionals wearing type IIR fluid resistant surgical masks
  Interventions: Behavioral: face masks

INTERVENTIONS:
Behavioral: face masks — wearing face masks

SUMMARY:
aim of this research is to evaluate the effects of FFP2/N95 masks on peripheral oxygen saturation and pulse rate in dental professionals

ELIGIBILITY:
Inclusion Criteria:

* dental professionals

Exclusion Criteria:

* subjects not signing informed consent
* subjects unable to wear facemasks due to underlying conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all kind of dental professionals
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
change in peripheral oxygen saturation using FFP2/N95 masks | before wearing face mask, after 30 minutes, after 1 hour, at the end of the clinical activity after 4-5 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Universitario A. Gemelli, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: Undecided